CLINICAL TRIAL: NCT05479929
Title: Work of Breathing Assessment in Triage Scale
Status: Active, not recruiting | Type: Observational
Sponsor: CHRISTUS Health (Other)
Responsible Party: Principal Investigator, Peter Richman, MD, Professor, CHRISTUS Health
Other Study IDs: 2020-195
Record Dates: First submitted 2022-07-21; First posted 2022-07-29 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Shortness of Breath; Respiratory Symptoms; Cough; Difficulty Breathing; Hypoxemia
Keywords: Emergency Room; Respiratory Assessment; Work of Breathing
MeSH Terms: conditions — Dyspnea; Signs and Symptoms, Respiratory; Cough; Hypoxia; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Respiratory Symptoms: The Canadian Triage Assessment Scale (CTAS) will be assessed via patient survey form and electronic chart review.
  Interventions: Other: Canadian Triage Assessment Scale (CTAS)

INTERVENTIONS:
Other: Canadian Triage Assessment Scale (CTAS) — The CTAS incorporates work of breathing into a subjective measurement in its assessment of patients and triaged.

SUMMARY:
The proposed research study will be a prospective observational study designed to validate the Canadian Triage Assessment Scale (CTAS) in regard to work of breathing in patients in the emergency department. The investigators will assess inter-rater agreement between nurses & emergency physicians for assessment of work of breathing.

DETAILED DESCRIPTION:
Investigators will enroll a convenience sample of consenting patients who present to the emergency department with a chief complaint related to respiratory symptoms, including shortness of breath, cough, difficulty breathing, hypoxemia, or any other respiratory related complaint.

Following consent and in a blinded fashion, the nurse & emergency physician will be asked to evaluate the patient's work of breathing into three subjective categories: mild, moderate, or severe. The two evaluators will not be aware of the others evaluation of the patient. Evaluators will also be asked to predict the patients likely need for intervention & disposition.

Subsequently, investigators will perform a chart review to determine the patient's clinical interventions, outcomes, and dispositions, and evaluate the assessment of the patients work of breathing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age of older
* Presenting to the emergency department with a chief complaint of any type of respiratory symptom.

Exclusion Criteria:

* Under 18 years of age
* Refusal to consent to study
* Incarcerated patients
* Pregnant patients
* Unable to complete survey due to clinical instability, severe pain, or disorientation determined by a study physician.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study subjects include any adult patients who present to the emergency department at Christus Spohn Hospital - Shoreline
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Inter-rater agreement between nurses and emergency physicians for the respiratory component of the Canadian Assessment Scale (CTAS) | 24 months
  The CTAS is utilized to qualitatively define work of breathing as severe, moderate, or mild. Kappa will be calculated to assess inter-rater reliability

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Durand, DO, Principal Investigator — CHRISTUS Health
Locations (1):
- CHRISTUS Spohn Hospital, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The Principal Investigator may want to pursue other opportunities with collaborators and sponsors.
Supporting Information: Study Protocol, ICF
Time Frame: 24 months

REFERENCES:
- [Background] Rui P, Kang K, Albert M. National Hospital Ambulatory Medical Care Survey: 2013 Emergency Department Summary Tables. Available from: http://www.cdc.gov/nchs/data/ahcd/nhamcs_emergency/2013_ed_web_tables.pdf.
- [Background] Hutchinson A, Pickering A, Williams P, Bland JM, Johnson MJ. Breathlessness and presentation to the emergency department: a survey and clinical record review. BMC Pulm Med. 2017 Mar 20;17(1):53. doi: 10.1186/s12890-017-0396-4. PMID 28320369
- [Background] Murray M, Bullard M, Grafstein E; CTAS Natioanal Working Group; CEDIS National Working Group. Revisions to the Canadian Emergency Department Triage and Acuity Scale implementation guidelines. CJEM. 2004 Nov;6(6):421-7. No abstract available. PMID 17378961
- [Background] Horeczko T, Enriquez B, McGrath NE, Gausche-Hill M, Lewis RJ. The Pediatric Assessment Triangle: accuracy of its application by nurses in the triage of children. J Emerg Nurs. 2013 Mar;39(2):182-9. doi: 10.1016/j.jen.2011.12.020. Epub 2012 Jul 24. PMID 22831826
- [Background] Jimenez JG, Murray MJ, Beveridge R, Pons JP, Cortes EA, Garrigos JB, Ferre MB. Implementation of the Canadian Emergency Department Triage and Acuity Scale (CTAS) in the Principality of Andorra: Can triage parameters serve as emergency department quality indicators? CJEM. 2003 Sep;5(5):315-22. PMID 17466139
- [Background] Alquraini M, Awad E, Hijazi R. Reliability of Canadian Emergency Department Triage and Acuity Scale (CTAS) in Saudi Arabia. Int J Emerg Med. 2015 Dec;8(1):80. doi: 10.1186/s12245-015-0080-5. Epub 2015 Aug 7. PMID 26251308
- [Background] Paniagua N, Elosegi A, Duo I, Fernandez A, Mojica E, Martinez-Indart L, Mintegi S, Benito J. Initial Asthma Severity Assessment Tools as Predictors of Hospitalization. J Emerg Med. 2017 Jul;53(1):10-17. doi: 10.1016/j.jemermed.2017.03.021. Epub 2017 Apr 14. PMID 28416251
- [Background] Roussos C, Koutsoukou A. Respiratory failure. Eur Respir J Suppl. 2003 Nov;47:3s-14s. doi: 10.1183/09031936.03.00038503. PMID 14621112
- [Background] Beveridge R, Ducharme J, Janes L, Beaulieu S, Walter S. Reliability of the Canadian emergency department triage and acuity scale: interrater agreement. Ann Emerg Med. 1999 Aug;34(2):155-9. doi: 10.1016/s0196-0644(99)70223-4. PMID 10424915